CLINICAL TRIAL: NCT05166109
Title: A Phase II Pilot Trial of Vamorolone vs. Placebo for the Treatment of Becker Muscular Dystrophy
Brief Title: A Study to Assess Vamorolone in Becker Muscular Dystrophy (BMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ReveraGen BioPharma, Inc. (Industry)
Collaborators: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VBP15-BMD-001; 1R01FD007284-01 (FDA)
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-12

CONDITIONS: Becker Muscular Dystrophy
Keywords: Becker Muscular Dystrophy; Duchenne Muscular Dystrophy; Duchenne and Becker Muscular Dystrophy; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — VBP15 compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vamorolone 500mg/day [250mg if <50kg body weight] (Experimental): Subjects will be randomized to one of two treatment groups in a 1:2 ratio (placebo:vamorolone).
  Interventions: Drug: Vamorolone
- Placebo (Placebo Comparator): Subjects will be randomized to one of two treatment groups in a 1:2 ratio (placebo:vamorolone).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vamorolone — Vamorolone 4.0% wt/wt oral suspension will be administered for the duration of the study.
  Other Names: VBP15
  Arms: Vamorolone 500mg/day [250mg if <50kg body weight]
Drug: Placebo — Placebo to Vamorolone 4.0% wt/wt oral suspension will be administered for the duration of the study.
  Other Names: Placebo to vamorolone
  Arms: Placebo

SUMMARY:
This Phase II pilot study is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, PD, and exploratory clinical efficacy of vamorolone 500mg (250mg for body weight <50 kg) daily administered orally compared to placebo over a treatment period of 24 weeks in males with BMD.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
This Phase II pilot study is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, PD, and exploratory clinical efficacy of vamorolone 500mg (250mg for body weight <50 kg) daily administered orally compared to placebo over a treatment period of 24 weeks in males with BMD.

The study is comprised of a Pretreatment Screening Period of up to 5 weeks duration (unless extended to accommodate varicella vaccination), a 1-day Pretreatment Baseline Period, a 24-week Treatment Period, and a 4-week Dose-tapering Period (for subjects not continuing directly with further vamorolone treatment). Subjects will be enrolled into this study at the time written informed consent is given, and administered study medication only after completion of all Pretreatment Screening assessments to confirm eligibility.

Subjects will be assessed for safety, tolerability, PK, PD, and effect on physical functioning at scheduled visits throughout the study. Screening assessments will be performed prior to baseline assessments on Day -1 and first administration of study medication on Day 1.

After completion of Screening and Baseline assessments, subjects will return to the study clinic on Day 1 for safety, PK and PD assessments prior to administration of the first dose of study medication. Additional on-site study visits will occur at Week 4, Week 12, and Week 24. Adverse events, including serious adverse events (SAEs), and concomitant medications will be recorded throughout the study. A Data and Safety Monitoring Board (DSMB) will review SAEs and other pertinent safety data at regular intervals during the study, and make recommendations to the Sponsor and Study Team regarding study conduct.

Subject diaries will be dispensed at the Day 1, Week 12, and Week 24 (for subjects participating in the Dose-tapering Period) Visits to record AEs, changes to concomitant medications taken during the study, and any missed or incomplete doses of study medication.

The scheduled Week 12 and Week 24 assessments may be performed over a 2-day period, if necessary, to facilitate scheduling.

Subjects who complete the VBP15-BMD-001 study assessments through the Week 24 Visit may be given the opportunity to continue to receive vamorolone as part of an expanded access or compassionate use program.

Subjects who complete the VBP15-BMD-001 study and will enroll directly into an expanded access or compassionate use program to continue vamorolone treatment will be discharged from the VBP15-BMD-001 study following completion of all Week 24 assessments. Subjects who will not continue vamorolone treatment in the expanded access or compassionate use program will have their study medication dose tapered during a 4-week Dose-tapering Period to taper study medication prior to discharge from the study. For these subjects, site study staff will contact the subject or parent(s)/guardian(s) by telephone at Week 26 to ensure that the dose tapering is proceeding according to protocol, to assess potential signs or symptoms of adrenal suppression, and to address any questions the subject or parent(s)/guardian(s) may have.

In the event that any clinical or laboratory parameters remain abnormal at the time of discharge from the study, the subject will be followed medically, as clinically indicated.

Any subject who discontinues the study prior to the Week 24 Visit should return to the study unit for scheduled Week 24 assessments at the time of early withdrawal and a Week 28 Visit following the taper, whenever possible, assuming the subject has not withdrawn consent. Any subject who withdraws early from the study after study medication dosing has begun should undergo dose-tapering following early completion of the Week 24 assessments and a Week 28 Visit following the taper.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or Subject's parent(s) or legal guardian (s) has (have) provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization, where applicable, prior to any study-related procedures;
2. Subject is a male and has a confirmed diagnosis of Becker dystrophy as defined as:

   1. Identifiable mutation within the DMD gene (deletion/duplication of one or more exons), where reading frame can be predicted as 'in-frame', and clinical picture consistent with Becker dystrophy, OR
   2. Complete dystrophin gene sequencing showing an alteration (small mutation, duplication, other) that is expected to allow production of an internally deleted dystrophin protein, with a typical clinical picture of Becker dystrophy;
3. Subject is ≥ 18 years of age and <65 years of age at time of informed consent;
4. Subject is able to perform the timed run/walk 10 meters assessment (TTRW) in ≤ 30 sec at screening; assistive devices, cane or walker, are allowed.
5. Subject has an NSAA score ≤ 32 at screening.
6. Clinical laboratory test results are within the normal range at the Screening Visit, or if abnormal, are not clinically significant, in the opinion of the Investigator. (Note: Serum gamma glutamyl transferase [GGT], creatinine, and total bilirubin all must be ≤ upper limit of the normal range at the Screening Visit). While AST and ALT can be elevated due to disease of muscle or liver, the study PI will review any increases of AST or ALT. If above upper limit of normal (ULN), then study PI will assess whether the increases are likely of muscle origin to determine inclusion.
7. Subject has not received oral glucocorticoids or other oral immunosuppressive agents for at least 3 months prior to first administration of study medication. [Note: Inhaled and/or topical glucocorticoids are permitted if last use is at least 4 weeks prior to first administration of study medication or if administered at stable dose beginning at least 4 weeks prior to first administration of study medication and anticipated to be used at the stable dose regimen for the duration of the study];
8. Subject has evidence of chicken pox immunity as determined by:

   1. Presence of IgG antibodies to varicella, as documented by a positive test result from the local laboratory from blood collected during the Screening Period; OR
   2. Documentation, provided at the Screening Visit, that the subject has received 2 doses of varicella vaccine, with or without serologic evidence of immunity, with the second of the 2 immunizations given at least 14 days prior to first administration of study medication;
9. Subject is willing and able to comply with scheduled visits, study medication administration plan, and study procedures.
10. Subject agrees to use barrier contraception methods during his participation in this study and for 30 days after the tapering dose is completed.

Exclusion Criteria:

1. Subject has current or history of major renal or hepatic impairment, uncontrolled diabetes mellitus (defined as a diagnosis of diabetes with random glucose more than 1.5x ULN at screening and the patient has symptoms of polyuria or polydipsia) or immunosuppression;
2. Subject has current or history of chronic systemic fungal or viral infections;
3. Subject has had an acute illness within 4 weeks prior to the first dose of study medication
4. Subject has used mineralocorticoid receptor agents, such as spironolactone, eplerenone, canrenone (canrenoate potassium), prorenone (prorenoate potassium), or mexrenone (mexrenoate potassium) within 4 weeks prior to administration of study medication;
5. Subject has evidence of symptomatic cardiomyopathy [Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary unless cardiac ejection fraction is less than 40%];
6. Subject has an allergy or hypersensitivity to the study medication or to any of its constituents;
7. Subject has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the Investigator;
8. Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator;
9. Subject is taking (or has taken within 4 weeks prior to first dose of study medication) herbal remedies and supplements which can impact muscle strength and function (e.g., Co-enzyme Q10, creatine, etc);
10. Subject has been administered a live attenuated vaccine within 14 days prior to the first dose of study medication;
11. Subject is currently taking any other investigational drug or has taken any other investigational drug within 3 months prior to first dose of study medication; or
12. Subject has previously been enrolled in the VBP15-BMD-001 study or any other vamorolone study.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Safety as measured by Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) by system organ class (SOC and PT) | 24 weeks
  Clinical AEs and clinical laboratory AEs will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, dated June 14, 2010.
  Dose-limiting toxicities will be defined as follows:
  1. The presence of a CTCAE Grade ≥ 3 AE, considered to be probably or definitely related to study drug
  2. The presence of a CTCAE Grade ≥ 3 clinical laboratory AE considered to be probably or definitely related to study drug
  3. Deterioration of the muscle condition, unexpected for the natural course of BMD and without other clear cause
Safety as measured by Sitting Blood Pressure | Day 1, Week 4, Week 12, Week 24, Week 28
  Change in Sitting Blood Pressure from baseline to each of the scheduled on-treatment and post-treatment assessment time points for each treatment group.
Safety as measured by Heart Rate | Day 1, Week 4, Week 12, Week 24, Week 28
  Change in Heart Rate from baseline to each of the scheduled on-treatment and post-treatment assessment time points for each treatment group.
Safety as measured by Respiratory Rate | Day 1, Week 4, Week 12, Week 24, Week 28
  Change in Respiratory Rate from baseline to each of the scheduled on-treatment and post-treatment assessment time points for each treatment group.
Safety as measured by Body Temperature | Day 1, Week 4, Week 12, Week 24, Week 28
  Change in Body Temperature from baseline to each of the scheduled on-treatment and post-treatment assessment time points for each treatment group.
Safety as measured by Body Weight | Week 12, Week 24, Week 28
  Change in Body Weight from baseline to each of the scheduled on-treatment and post-treatment assessment time points for each treatment group.
Safety as measured by Height | Week 12, Week 24, Week 28
  Change in Height from screening to each of the scheduled on-treatment and post-treatment assessment time points for each treatment group.
Safety: concentration of blood laboratory biomarkers as assessed by standardized clinical laboratory reference ranges | Week 4, Week 12, Week 24
  Blood biomarkers are White Blood cells (WBCs), Red Blood Cells, (RBCs), hemoglobin, Platelets, Sodium, Potassium, Chloride, Calcium, Blood Urea Nitrogen (BUN), Creatinine, Total Protein, Albumin, Total Bilirubin, Glucose, Alkaline Phosphatase (ALP), Gamma Glutamyl Transferase (GGT), Glutamate Dehydrogenase (GLDH), Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Creatine kinase (CK), Bicarbonate, Triglycerides, Total cholesterol, Low Density Lipoprotein (LDL) and High density Lipoprotein (HDL). Change from baseline to each of the scheduled on treatment and post-treatment time points will be assessed.
Safety: concentration of urine laboratory biomarkers as measured by dipstick and microscopic analysis | Week 4, Week 12, Week 24
  Urine biomarkers are protein, glucose, ketones, leukocyte esterase, White Blood Cells (WBCs), Red Blood Cells, (RBCs) and bacteria. Change from baseline to each of the scheduled on treatment and post-treatment time points will be assessed.
Safety as measured by 12-lead ECG | Week 12, Week 24
  12-lead ECG as recorded after subject has rested quietly in a supine position for at least 5 minutes. ECG components are QRS duration, PR interval, QT interval and QTc interval. Change from baseline to each of the scheduled on-treatment and post-treatment assessment time points.
Tolerability as measured by incidence of Premature Discontinuation | 24 weeks
  Premature Discontinuation of study treatment due to adverse event.

SECONDARY OUTCOMES:
Pharmacokinetics as measured by AUCinf | Day 1
  Blood will be collected from all subjects at the Day 1 Visit, at 1, 2 and 3 hours post-dose, for vamorolone PK analysis
Safety as measured by serum concentration of osteocalcin | Week 24
  Change from baseline to Week 24 will be assessed for each treatment group.
Safety as measured by serum concentration of hemoglobin A1c (HbA1c) | Week 24
  Change from baseline to Week 24 will be assessed for each treatment group.
Safety as measured by fasting serum concentration of glucose | Week 12, Week 24
  Change from baseline to each of the scheduled study assessment time points for each treatment group.
Safety as measured by fasting serum concentration of insulin | Week 12, Week 24
  Change from baseline to each of the scheduled study assessment time points for each treatment group.
Efficacy as measured by concentration of serum pharmacodynamic biomarkers | Week 12, Week 24
  CD23 (also known as Fc epsilon RII) and Macrophage Derived Chemokine (MDC) and concentration from baseline to Week 24.
Safety as measured by concentration of Salivary Cortisol | Day 1, Week 12, Week 24
  First-in-morning salivary cortisol levels will be measured. Cortisol measures falling below 3.6 µg/dL (or 100 nM) will be considered to be indicative of the development of adrenal suppression. Cortisol will be assessed for each treatment group.

OTHER OUTCOMES:
Efficacy as measured by Time to Run/Walk Test (TTRW) | Week 12, Week 24
  Change from baseline to each of the scheduled assessment time points for each treatment group.
Efficacy as measured by North Star Ambulatory Assessment (NSAA) score | Week 12, Week 24
  Change from baseline to each of the scheduled assessment time points for each treatment group.
Tolerability as measured by NeuroQOL score | 24 weeks
  Participants or participants' parent(s)/legal guardian(s) will be asked to complete the NeuroQOL scales for fatigue, upper and lower extremities function and sleep. Change from baseline to 24 weeks will be assessed by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Clemens, M.D., Study Chair — University of Pittsburgh
Locations (2):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States
- Azienda Ospedale Universita Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffman EP, Schwartz BD, Mengle-Gaw LJ, Smith EC, Castro D, Mah JK, McDonald CM, Kuntz NL, Finkel RS, Guglieri M, Bushby K, Tulinius M, Nevo Y, Ryan MM, Webster R, Smith AL, Morgenroth LP, Arrieta A, Shimony M, Siener C, Jaros M, Shale P, McCall JM, Nagaraju K, van den Anker J, Conklin LS, Cnaan A, Gordish-Dressman H, Damsker JM, Clemens PR; Cooperative International Neuromuscular Research Group. Vamorolone trial in Duchenne muscular dystrophy shows dose-related improvement of muscle function. Neurology. 2019 Sep 24;93(13):e1312-e1323. doi: 10.1212/WNL.0000000000008168. Epub 2019 Aug 26. PMID 31451516
- [Background] Smith EC, Conklin LS, Hoffman EP, Clemens PR, Mah JK, Finkel RS, Guglieri M, Tulinius M, Nevo Y, Ryan MM, Webster R, Castro D, Kuntz NL, Kerchner L, Morgenroth LP, Arrieta A, Shimony M, Jaros M, Shale P, Gordish-Dressman H, Hagerty L, Dang UJ, Damsker JM, Schwartz BD, Mengle-Gaw LJ, McDonald CM; CINRG VBP15 and DNHS Investigators. Efficacy and safety of vamorolone in Duchenne muscular dystrophy: An 18-month interim analysis of a non-randomized open-label extension study. PLoS Med. 2020 Sep 21;17(9):e1003222. doi: 10.1371/journal.pmed.1003222. eCollection 2020 Sep. PMID 32956407
- [Background] Heier CR, Yu Q, Fiorillo AA, Tully CB, Tucker A, Mazala DA, Uaesoontrachoon K, Srinivassane S, Damsker JM, Hoffman EP, Nagaraju K, Spurney CF. Vamorolone targets dual nuclear receptors to treat inflammation and dystrophic cardiomyopathy. Life Sci Alliance. 2019 Feb 11;2(1):e201800186. doi: 10.26508/lsa.201800186. Print 2019 Feb. PMID 30745312
- [Background] Mavroudis PD, van den Anker J, Conklin LS, Damsker JM, Hoffman EP, Nagaraju K, Clemens PR, Jusko WJ. Population Pharmacokinetics of Vamorolone (VBP15) in Healthy Men and Boys With Duchenne Muscular Dystrophy. J Clin Pharmacol. 2019 Jul;59(7):979-988. doi: 10.1002/jcph.1388. Epub 2019 Feb 11. PMID 30742306
- [Background] Damsker JM, Cornish MR, Kanneboyina P, Kanneboyina I, Yu Q, Lipson R, Phadke A, Knoblach SM, Panchapakesan K, Morales M, Fiorillo AA, Partridge T, Nagaraju K. Vamorolone, a dissociative steroidal compound, reduces collagen antibody-induced joint damage and inflammation when administered after disease onset. Inflamm Res. 2019 Nov;68(11):969-980. doi: 10.1007/s00011-019-01279-z. Epub 2019 Aug 24. PMID 31446438
- [Background] Akkad H, Cacciani N, Llano-Diez M, Corpeno Kalamgi R, Tchkonia T, Kirkland JL, Larsson L. Vamorolone treatment improves skeletal muscle outcome in a critical illness myopathy rat model. Acta Physiol (Oxf). 2019 Feb;225(2):e13172. doi: 10.1111/apha.13172. Epub 2018 Sep 6. PMID 30120816
- [Background] Li X, Conklin LS, van den Anker J, Hoffman EP, Clemens PR, Jusko WJ. Exposure-Response Analysis of Vamorolone (VBP15) in Boys With Duchenne Muscular Dystrophy. J Clin Pharmacol. 2020 Oct;60(10):1385-1396. doi: 10.1002/jcph.1632. Epub 2020 May 20. PMID 32434278
- [Background] Hoffman EP, Riddle V, Siegler MA, Dickerson D, Backonja M, Kramer WG, Nagaraju K, Gordish-Dressman H, Damsker JM, McCall JM. Phase 1 trial of vamorolone, a first-in-class steroid, shows improvements in side effects via biomarkers bridged to clinical outcomes. Steroids. 2018 Jun;134:43-52. doi: 10.1016/j.steroids.2018.02.010. Epub 2018 Mar 8. PMID 29524454
- [Background] Almeida LEF, Damsker JM, Albani S, Afsar N, Kamimura S, Pratt D, Kleiner DE, Quezado M, Gordish-Dressman H, Quezado ZMN. The corticosteroid compounds prednisolone and vamorolone do not alter the nociception phenotype and exacerbate liver injury in sickle cell mice. Sci Rep. 2018 Apr 17;8(1):6081. doi: 10.1038/s41598-018-24274-6. PMID 29666400
- [Background] Wells E, Kambhampati M, Damsker JM, Gordish-Dressman H, Yadavilli S, Becher OJ, Gittens J, Stampar M, Packer RJ, Nazarian J. Vamorolone, a dissociative steroidal compound, reduces pro-inflammatory cytokine expression in glioma cells and increases activity and survival in a murine model of cortical tumor. Oncotarget. 2017 Feb 7;8(6):9366-9374. doi: 10.18632/oncotarget.14070. PMID 28030841
- [Background] Liu X, Wang Y, Gutierrez JS, Damsker JM, Nagaraju K, Hoffman EP, Ortlund EA. Disruption of a key ligand-H-bond network drives dissociative properties in vamorolone for Duchenne muscular dystrophy treatment. Proc Natl Acad Sci U S A. 2020 Sep 29;117(39):24285-24293. doi: 10.1073/pnas.2006890117. Epub 2020 Sep 11. PMID 32917814
- [Background] Conklin LS, Damsker JM, Hoffman EP, Jusko WJ, Mavroudis PD, Schwartz BD, Mengle-Gaw LJ, Smith EC, Mah JK, Guglieri M, Nevo Y, Kuntz N, McDonald CM, Tulinius M, Ryan MM, Webster R, Castro D, Finkel RS, Smith AL, Morgenroth LP, Arrieta A, Shimony M, Jaros M, Shale P, McCall JM, Hathout Y, Nagaraju K, van den Anker J, Ward LM, Ahmet A, Cornish MR, Clemens PR. Phase IIa trial in Duchenne muscular dystrophy shows vamorolone is a first-in-class dissociative steroidal anti-inflammatory drug. Pharmacol Res. 2018 Oct;136:140-150. doi: 10.1016/j.phrs.2018.09.007. Epub 2018 Sep 13. PMID 30219580
- [Background] Fiorillo AA, Tully CB, Damsker JM, Nagaraju K, Hoffman EP, Heier CR. Muscle miRNAome shows suppression of chronic inflammatory miRNAs with both prednisone and vamorolone. Physiol Genomics. 2018 Sep 1;50(9):735-745. doi: 10.1152/physiolgenomics.00134.2017. Epub 2018 Jun 8. PMID 29883261
- [Background] Sreetama SC, Chandra G, Van der Meulen JH, Ahmad MM, Suzuki P, Bhuvanendran S, Nagaraju K, Hoffman EP, Jaiswal JK. Membrane Stabilization by Modified Steroid Offers a Potential Therapy for Muscular Dystrophy Due to Dysferlin Deficit. Mol Ther. 2018 Sep 5;26(9):2231-2242. doi: 10.1016/j.ymthe.2018.07.021. Epub 2018 Aug 27. PMID 30166241
- [Background] Dang UJ, Ziemba M, Clemens PR, Hathout Y, Conklin LS; CINRG Vamorolone 002/003 Investigators; Hoffman EP. Serum biomarkers associated with baseline clinical severity in young steroid-naive Duchenne muscular dystrophy boys. Hum Mol Genet. 2020 Aug 29;29(15):2481-2495. doi: 10.1093/hmg/ddaa132. PMID 32592467
- [Background] Ziemba M, Barkhouse M, Uaesoontrachoon K, Giri M, Hathout Y, Dang UJ, Gordish-Dressman H, Nagaraju K, Hoffman EP. Biomarker-focused multi-drug combination therapy and repurposing trial in mdx mice. PLoS One. 2021 Feb 22;16(2):e0246507. doi: 10.1371/journal.pone.0246507. eCollection 2021. PMID 33617542
- [Background] Dadgar S, Wang Z, Johnston H, Kesari A, Nagaraju K, Chen YW, Hill DA, Partridge TA, Giri M, Freishtat RJ, Nazarian J, Xuan J, Wang Y, Hoffman EP. Asynchronous remodeling is a driver of failed regeneration in Duchenne muscular dystrophy. J Cell Biol. 2014 Oct 13;207(1):139-58. doi: 10.1083/jcb.201402079. PMID 25313409
- [Background] Heier CR, Damsker JM, Yu Q, Dillingham BC, Huynh T, Van der Meulen JH, Sali A, Miller BK, Phadke A, Scheffer L, Quinn J, Tatem K, Jordan S, Dadgar S, Rodriguez OC, Albanese C, Calhoun M, Gordish-Dressman H, Jaiswal JK, Connor EM, McCall JM, Hoffman EP, Reeves EK, Nagaraju K. VBP15, a novel anti-inflammatory and membrane-stabilizer, improves muscular dystrophy without side effects. EMBO Mol Med. 2013 Oct;5(10):1569-85. doi: 10.1002/emmm.201302621. Epub 2013 Sep 9. PMID 24014378
- [Background] Damsker JM, Dillingham BC, Rose MC, Balsley MA, Heier CR, Watson AM, Stemmy EJ, Jurjus RA, Huynh T, Tatem K, Uaesoontrachoon K, Berry DM, Benton AS, Freishtat RJ, Hoffman EP, McCall JM, Gordish-Dressman H, Constant SL, Reeves EK, Nagaraju K. VBP15, a glucocorticoid analogue, is effective at reducing allergic lung inflammation in mice. PLoS One. 2013 May 7;8(5):e63871. doi: 10.1371/journal.pone.0063871. Print 2013. PMID 23667681
- [Background] Freishtat RJ, Nino G, Tsegaye Y, Alcala SE, Benton AS, Watson AM, Reeves EK, Haider SK, Damsker JM. Pharmacologically-induced mitotic synchrony in airway epithelial cells as a mechanism of action of anti-inflammatory drugs. Respir Res. 2015 Oct 29;16:132. doi: 10.1186/s12931-015-0293-4. PMID 26511361
- [Background] Dillingham BC, Knoblach SM, Many GM, Harmon BT, Mullen AM, Heier CR, Bello L, McCall JM, Hoffman EP, Connor EM, Nagaraju K, Reeves EKM, Damsker JM. VBP15, a novel anti-inflammatory, is effective at reducing the severity of murine experimental autoimmune encephalomyelitis. Cell Mol Neurobiol. 2015 Apr;35(3):377-387. doi: 10.1007/s10571-014-0133-y. Epub 2014 Nov 13. PMID 25392236
- [Background] Garvin LM, Chen Y, Damsker JM, Rose MC. A novel dissociative steroid VBP15 reduces MUC5AC gene expression in airway epithelial cells but lacks the GRE mediated transcriptional properties of dexamethasone. Pulm Pharmacol Ther. 2016 Jun;38:17-26. doi: 10.1016/j.pupt.2016.04.004. Epub 2016 Apr 29. PMID 27133900
- [Background] Damsker JM, Conklin LS, Sadri S, Dillingham BC, Panchapakesan K, Heier CR, McCall JM, Sandler AD. VBP15, a novel dissociative steroid compound, reduces NFkappaB-induced expression of inflammatory cytokines in vitro and symptoms of murine trinitrobenzene sulfonic acid-induced colitis. Inflamm Res. 2016 Sep;65(9):737-43. doi: 10.1007/s00011-016-0956-8. Epub 2016 Jun 3. PMID 27261270